CLINICAL TRIAL: NCT06886542
Title: Comparison of the Effectiveness of Single and Dual Task Training Applied to Individuals With Knee Meniscus Lesion: A Randomized Controlled, Single-Blind Study
Brief Title: Comparison of the Effectiveness of Single and Dual Task Training Applied to Individuals With Knee Meniscus Lesion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26.12.24/ 10-1059
Record Dates: First submitted 2025-03-07; First posted 2025-03-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-03

CONDITIONS: Meniscus Lesion
Keywords: knee meniscus lesion; dual task training

STUDY DESIGN:
Intervention Model Description: Parallel Assignment dual parallel group design
Who Masked: Outcomes Assessor
Masking Description: The evaluation of the patients will be carried out by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Patients in this group are the group to which dual task training and conventional physiotherapy will be applied
  Interventions: Other: Dual task training; Other: Conventional physiotherapy
- Control group (Active Comparator): Patients in this group are the group to which single task training and conventional physiotherapy will be applied.
  Interventions: Other: Single task training; Other: Conventional physiotherapy

INTERVENTIONS:
Other: Dual task training — Dual task training is based on the simultaneous maintenance of motor-motor or cognitive-motor performance. The exercises given in single task training will be applied by combining them with cognitive and motor cognitive tasks.
  Arms: Treatment group
Other: Single task training — Single task training is a training approach that aims to improve the performance of individuals by focusing on only one task at a time.
  Arms: Control group
Other: Conventional physiotherapy — Range of motion, stretching, resistance exercises, isometric exercise, Before the treatment, a Hotpack will be applied to warm up the muscles, increase flexibility and improve performance. After exercise, transcutaneous electrical stimulation (TENS) will be used to relieve pain, reduce muscle tension and provide faster recovery.

SUMMARY:
The main function of the meniscus is to transfer and distribute femoral pressure to the tibia. Treatment of meniscus tears is divided into conservative and surgical treatment. The most preferred methods for patients with meniscus lesions include meniscectomy and exercise therapy. The anterior and posterior horns of the meniscus contain numerous mechanoreceptors, including Ruffini endings (slow adapting) and Pacinian corpuscles (fast adapting), which provide information about the position and movement of the joint. Reduced proprioception due to mechanoreceptor damage from meniscus tears may be associated with decreased postural stability, as sensory information associated with a patient's conscious perception of joint movement through mechanoreceptors in the meniscus may contribute to postural stability.

Dual task is based on the simultaneous maintenance of motor-motor or cognitive-motor performance. Dual tasking is used to evaluate the simultaneous performance of a postural task and a motor or cognitive task to examine the interaction or effect of the secondary task on primary task performance. In a purposeful movement, it is necessary to have the ability to adapt to overcome environmental loads and achieve the goal. This also involves performing a cognitive task simultaneously while performing a motor task. In knee meniscus lesions, knee joint position sense and sensory input decrease, walking speed decreases, and attention devoted to walking increases.

DETAILED DESCRIPTION:
Complex movement formation needs to be restructured as a result of sensory and motor disorders. With the loss of movement organization, postural control becomes vulnerable to cognitive attention elements and additional motor tasks. While physical disability creates a burden for the individual and society, it also has a negative impact on executive functions. Robust cognitive processes are essential when performing complex motor tasks and ensuring stable walking. Because the dependence on cognitive resources increases to compensate for the loss of control in postural stability and balance. Although walking and balance are considered to be automatic tasks, performance decreases when processing capacity is exceeded by a simultaneous task. In dual task studies, it has been reported that there is an increase in step time and a decrease in step length due to the increase in the single and double support phases of walking. This situation has been interpreted as a strategy developed to maintain balance in dual task conditions. With the dual task training to be applied to these individuals, it is aimed to ensure that motor control, balance, and the complex movements they encounter in daily life activities can be maintained in balance while walking.

ELIGIBILITY:
Inclusion Criteria:

* 40 to 65 years old
* According to magnetic resonance imaging (MRI) results, there is a maximum of Grade 2 degenerative bilateral meniscus tear
* Having a Standardized Mini Mental Test score of 24 and above
* Volunteering
* Know how to read and write
* Not having vision or hearing problems that cannot be corrected with a device
* Being able to walk independently in society

Exclusion Criteria:

* Not meeting the inclusion criteria
* Having compliance issues or emotional and cognitive problems that will prevent participation in the assessments and clinical practices to be used in the study
* Having problems participating in exercises or follow-ups
* Having had surgery related to the lower extremity
* Having a neuromuscular disease
* Having a history of systemic inflammatory joint disease
* Having a rheumatic disease
* Having an additional pathology in the knee
* Receiving additional treatment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-17 (Estimated); Primary Completion 2026-08-17 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance | Change from baseline at 8 weeks treatment program and two months after.
  The Modified Four Square Step Test will be used in the dynamic balance assessment.The test involves changing direction while taking steps forward, backward, and sideways. Individuals will be asked to stand in square number 1 and face square number 2. The movement will be started and they will be asked to step into squares number 2,3,4,1,4,3,2,1 in order. First, they will take a turn clockwise and then counterclockwise. Two measurements will be made and the average value will be recorded in seconds. The test will be repeated with single task, cognitive dual task and motor dual task.
Static Balance | Change from baseline at 8 weeks treatment program and two months after.
  Static balance will be assessed with a one-leg standing test.The test starts when one foot leaves the ground and ends when it touches the ground again, in case of excessive oscillation or jumping with the foot on the ground. The person is asked to stand on one leg for as long as possible. The test is terminated when 30 seconds are reached. The test will be applied to bilateral lower extremities with single task, cognitive dual task, and motor dual task.
Gait Evaluation | Change from baseline at 8 weeks treatment program and two months after.
  A 10-meter walking test will be used to evaluate individuals' walking. Two measurements will be made and the average value will be recorded in seconds. The test will be repeated with single task, cognitive dual task and motor dual task.
Assessment of Functional Mobility | Change from baseline at 8 weeks treatment program and two months after.
  The Timed Up and Go Test will be used to assess functional mobility. In this test, the individual is asked to stand up while sitting in a chair with armrests and no wheels with the command 'Start', walk at his/her normal pace on a flat surface to a colored tape that was previously attached 3 meters away, then turn around and walk back to the chair and sit down again. The test will be repeated twice and the average time will be recorded in seconds. The test will be repeated with a single task, a cognitive dual task and a motor dual task.
Joint Position Sense | Change from baseline at 8 weeks treatment program and two months after.
  Joint position sense is evaluated by the angular difference between a repeatedly determined target position and the estimated position, and this is called absolute angular error. 30° and 60° knee flexion will be determined as target angles. A smartphone measurement application will be used for measurement. For the test position, individuals will be seated with their hips and knees at 90° flexion and their feet off the ground, and while the knee is slowly brought from 90° flexion to passive extension, individuals will be asked to perceive and learn this position by first stopping at 60° flexion angle for 5 seconds. Then, the individual will be asked to bring their knee to this target angle and the measurement will be made. The difference will be recorded as absolute angular error. The same process will be done for 30° flexion angle. Three repetitions will be requested for both positions and the averages will be calculated and recorded.

SECONDARY OUTCOMES:
Functional Capacity Assessment | Change from baseline at 8 weeks treatment program and two months after.
  The timed sit-to-stand test is a test used to measure muscular strength and endurance. The individual is asked to sit down and stand up as many times as possible in 30 seconds without support from a 43-45 cm high chair without armrests, with their feet shoulder-width apart, and the number reached is recorded.
Evaluation of the Functional Level of the Knee | Change from baseline at 8 weeks treatment program and two months after.
  The Western Ontario Meniscal Evaluation Tool (WOMET) will be used in this evaluation. This inventory includes 16 items representing the areas of influence of physical symptoms (nine items), sports/leisure/work/lifestyle (four items) and emotions (three items). A value between "0-10" is requested for each item. The score for each subgroup is obtained by dividing the marked values of the questions belonging to that section by the number of questions and multiplying by 10. The total score is obtained by adding all the scores, dividing by 16 and multiplying by 10.
Dual Task Assessment | Change from baseline at 8 weeks treatment program and two months after.
  The evaluation of dual task performance will be done with the Dual Task Evaluation Questionnaire. The Likert type survey consists of 10 questions. It includes the answers (4) very often, (3) often, (2) sometimes, (1) rarely and not applicable. The total score is calculated as the average value per question.
Pain level | Change from baseline at 8 weeks treatment program and two months after.
  Visual analog scale will be used to examine pain levels of participants. Individuals are presented with a line numbered evenly from 1 to 10 and asked to mark the point corresponding to their pain intensity. A higher score indicates that severity of pain increasing.
Muscle Strength Measurement | Change from baseline at 8 weeks treatment program and two months after.
  In this evaluation, a Lafayette brand digital hand dynamometer will be used. This device objectively shows the amount of force used in the muscle test. The knee extension force will be determined by placing the dynamometer distal to the tibia while the patient is in a sitting position and the knee is flexed at 65 degrees, and the patient will be asked to perform a maximal isometric contraction. The knee flexion force will be determined by placing the dynamometer distal to the tibia while the patient is in a prone position and the knee is flexed at 75 degrees, and the patient will be asked to perform a maximal isometric contraction. The measurement will be repeated 3 times and the highest value will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Rumeysa Reis Kul MSc, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Recep Tayyip Erdoğan University, Rize, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Indivudual participant data will be available to the responsible researcher.